CLINICAL TRIAL: NCT02980380
Title: Brain Computer Interface Based Communication in the Completely Locked-In State
Brief Title: Brain Computer Interface Complete locked-in State Communication
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, Dr. Ujwal Chaudhary, Principal Investigator, University Hospital Tuebingen
Other Study IDs: ALS BCI study
Record Dates: First submitted 2016-11-22; First posted 2016-12-02 (Estimated); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: Complete Locked-in State
Keywords: non-invasive brain computer interface; communication; amyotrophic lateral sclerosis; complete locked-in state
MeSH Terms: conditions — Communication; Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Locked-in and complete locked-in state patients: Amyotrophic lateral sclerosis patients in complete locked-in state as well as in transition from locked-in to complete locked-in state who have no means of communication.
  Interventions: Other: Non-invasive brain computer interface

INTERVENTIONS:
Other: Non-invasive brain computer interface — The hemodynamic change in the motor cortex of the CLIS patient will be recorded across many sessions spread over more than a year and will be used to train a classifier to predict the "yes" and "no" answering pattern of the CLIS patient. For patient who can still open their eyes but cannot use any other means of communication will control an EEG based BCI for communication.

SUMMARY:
Electroencephalography (EEG) and/or near-infrared spectroscopy (NIRS) based Brain computer interface for communication in patients without any means of communication.

DETAILED DESCRIPTION:
Amyotrophic lateral sclerosis is a progressive motor disease of unknown etiology resulting eventually in a complete paralysis of the motor system but affecting sensory or cognitive functions to a minor degree. There is no treatment available; patients have to decide to accept artificial respiration and feeding after the disease destroys respiratory and bulbar functions or to die of respiratory or related problems. If they opt for life and accept artificial respiration, the disease progresses until the patient loses control of the last muscular response, usually the eye muscles. If rudimentary voluntary control of at least one muscle is present the syndrome is called locked-in state (LIS); ultimately as the disease progresses most ALS patients lose the control of all muscles, the resulting condition is called completely locked-in state (CLIS). Patients in CLIS are unable to communicate with the external world because all assistive communication aids are based on some remaining motor control; hence there is a vital need for an assistive technology to help patients in CLIS to communicate needs and feelings to their family members/caregivers. Brain computer interface (BCI) represents a promising strategy to establish communication with paralyzed ALS patients, as it does not need muscle control. BCI research includes invasive (implantable electrodes on or in the neocortex) and noninvasive means (including electroencephalography (EEG), magnetoencephalography (MEG), functional magnetic resonance imaging (fMRI), and near-infrared spectroscopy (NIRS)) to record brain activity for conveying the user's intent to devices such as simple word-processing programs. Non-invasive methods have been utilized more frequently than invasive methods for people with disabilities (such as those with ALS).

For these conditions (LIS and CLIS) Brain-Computer-Interface were developed and tested extensively since the first publication of Birbaumer, 1999 of two LIS patients suffering from ALS. Patients select letters or words after learning self-regulation of the particular brain signal or by focusing their attention to the desired letter or a letter-matrix and the attention related brain potential selects the desired letter.

Different types of BCI based on EEG and/NIRS is under development to provide a means of communication to patients who have none.

ELIGIBILITY:
Inclusion Criteria:

* Amyotrophic lateral sclerosis patients without any eye movement

Exclusion Criteria:

* Amyotrophic lateral sclerosis patients with intact eye movement

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Amyotrophic lateral sclerosis patients in complete locked-in state without any eye movement
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2014-06 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Brain Computer Interface Based Communication in the Completely Locked-In State patients | 2 years
  fNIRS based BCI will be employed for communication in ALS patients in CLIS. The hemodynamic change in the motor cortex of the CLIS patient will be recorded and will be used for communication.

CONTACTS AND LOCATIONS:
Overall Officials: Niels Birbaumer, PhD, Principal Investigator — University Hospital Tuebingen
Locations (1):
- University of Tuebingen, Tübingen, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Undecided
Data will be made available to other researcher after publication of the study

REFERENCES:
- [Background] Birbaumer N. Breaking the silence: brain-computer interfaces (BCI) for communication and motor control. Psychophysiology. 2006 Nov;43(6):517-32. doi: 10.1111/j.1469-8986.2006.00456.x. PMID 17076808
- [Background] Birbaumer N, Ghanayim N, Hinterberger T, Iversen I, Kotchoubey B, Kubler A, Perelmouter J, Taub E, Flor H. A spelling device for the paralysed. Nature. 1999 Mar 25;398(6725):297-8. doi: 10.1038/18581. No abstract available. PMID 10192330
- [Background] Birbaumer N, Cohen LG. Brain-computer interfaces: communication and restoration of movement in paralysis. J Physiol. 2007 Mar 15;579(Pt 3):621-36. doi: 10.1113/jphysiol.2006.125633. Epub 2007 Jan 18. PMID 17234696
- [Background] Chaudhary U, Birbaumer N, Curado MR. Brain-machine interface (BMI) in paralysis. Ann Phys Rehabil Med. 2015 Feb;58(1):9-13. doi: 10.1016/j.rehab.2014.11.002. Epub 2015 Jan 8. PMID 25623294
- [Background] van Gerven M, Farquhar J, Schaefer R, Vlek R, Geuze J, Nijholt A, Ramsey N, Haselager P, Vuurpijl L, Gielen S, Desain P. The brain-computer interface cycle. J Neural Eng. 2009 Aug;6(4):041001. doi: 10.1088/1741-2560/6/4/041001. Epub 2009 Jul 22. PMID 19622847
- [Background] Farwell LA, Donchin E. Talking off the top of your head: toward a mental prosthesis utilizing event-related brain potentials. Electroencephalogr Clin Neurophysiol. 1988 Dec;70(6):510-23. doi: 10.1016/0013-4694(88)90149-6. PMID 2461285
- [Background] Kubler A, Birbaumer N. Brain-computer interfaces and communication in paralysis: extinction of goal directed thinking in completely paralysed patients? Clin Neurophysiol. 2008 Nov;119(11):2658-66. doi: 10.1016/j.clinph.2008.06.019. Epub 2008 Sep 27. PMID 18824406
- [Background] De Massari D, Ruf CA, Furdea A, Matuz T, van der Heiden L, Halder S, Silvoni S, Birbaumer N. Brain communication in the locked-in state. Brain. 2013 Jun;136(Pt 6):1989-2000. doi: 10.1093/brain/awt102. Epub 2013 Apr 26. PMID 23625062
- [Background] Gallegos-Ayala G, Furdea A, Takano K, Ruf CA, Flor H, Birbaumer N. Brain communication in a completely locked-in patient using bedside near-infrared spectroscopy. Neurology. 2014 May 27;82(21):1930-2. doi: 10.1212/WNL.0000000000000449. Epub 2014 Apr 30. PMID 24789862